CLINICAL TRIAL: NCT04334538
Title: Effect of an Alternative RUTF on Intestinal Permeability in Children With Severe Acute Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Project Peanut Butter, Sierra Leone (Unknown); Ministry of Health and Sanitation, Sierra Leone (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202003153
Record Dates: First submitted 2020-03-30; First posted 2020-04-06 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Malnutrition, Child
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S-RUTF (Active Comparator): Children will receive approximately 175 kcal/kg/d of standard ready to use therapeutic food which provides a full daily doses of vitamins and micronutrients. Caregivers will instruct caregivers to feed the supplement only to the enrolled child.
  Interventions: Dietary Supplement: S-RUTF
- oat-RUTF (Experimental): Children will receive approximately 175 kcal/kg/d of oat ready-to-use therapeutic food which provides a full daily doses of vitamins and micronutrients. Caregivers will instruct caregivers to feed the supplement only to the enrolled child.
  Interventions: Dietary Supplement: oat RUTF

INTERVENTIONS:
Dietary Supplement: S-RUTF — Children will receive approximately 175 kcal/kg/d of standard ready-to-use therapeutic food which provides a full daily doses of vitamins and micronutrients. Caregivers will instruct caregivers to feed the supplement only to the enrolled child.
  Arms: S-RUTF
Dietary Supplement: oat RUTF — Children will receive approximately 175 kcal/kg/d of oat ready-to-use therapeutic food which provides a full daily doses of vitamins and micronutrients. Caregivers will instruct caregivers to feed the supplement only to the enrolled child.
  Arms: oat-RUTF

SUMMARY:
Ready-to-use therapeutic food (RUTF) is the standard of care for the treatment of SAM. UNICEF requires that there be no oil separation in these products necessitating the use of emulsifiers. The effect of emulsifiers on gut health and integrity in children receiving an exclusive diet of RUTF is unknown. The PIs have recently completed a randomized, triple-blind, controlled, clinical equivalency trial in Sierra Leone comparing the alternative oat RUTF (oat-RUTF) to standard RUTF on recovery rates in children with SAM. This study demonstrated higher rates of recovery among children receiving the oat-RUTF. The investigators hypothesize that this benefit may be due to the lack of emulsifier in the oat-RUTF resulting in improved intestinal health.This research project is a double-blind, randomized, controlled clinical effectiveness trial comparing a novel RUTF containing oats and no emulsifier and standard RUTF on recovery from severe acute malnutrition (SAM) and effects on intestinal health. The trial will be conducted in up to 40 PHUs in Western Rural and Pujehun Districts where supplementary feeding programs (SFP) are not currently available.

ELIGIBILITY:
Inclusion Criteria:

* mid-upper arm circumference (MUAC) <11.5 cm

Exclusion Criteria:

* Children currently involved in another research trial or feeding program
* Children developmentally delayed
* have a chronic debilitating illness
* history of peanut or milk allergy

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 129 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
Change of % of lactose excreted between enrollment and 4 weeks after enrollment | at week 4 after enrollment
  %L measured in the urine relative to the amount ingested will be calculated for children in both groups. %L will be categorized as normal (<0.2%) and abnormal (>0.2)

SECONDARY OUTCOMES:
fecal 16S rRNA configuration after 4 weeks of feeding | after 4 weeks of feeding
  Multi amplicon rRNA characterization of flash frozen stool sample

CONTACTS AND LOCATIONS:
Locations (1):
- Project Peanut Butter, Pujehun, Sierra Leone

REFERENCES:
- [Derived] Hendrixson DT, Naskidashvili N, Stephenson KB, Laury ML, Koroma AS, Manary MJ. An Alternative Oat-Containing, Ready-To-Use, Therapeutic Food Does Not Alter Intestinal Permeability or the 16S Ribosomal RNA Fecal Microbiome Configuration Among Children With Severe Malnutrition in Sierra Leone: A Randomized Controlled Trial. J Nutr. 2023 Jan 14;152(12):2744-2753. doi: 10.1093/jn/nxac207. PMID 36055798